CLINICAL TRIAL: NCT05852977
Title: Study of Dengue in Patients With Autoimmune Diseases With or Without Immunosuppressive Treatment During the Epidemics of 2020 and 2021 in Reunion Island
Brief Title: Study of Dengue in Patients With Autoimmune Diseases During the Epidemics of 2020 and 2021 in Reunion Island
Acronym: MAIDEN
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/24
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is not known whether there is a different clinical profile of dengue in patients with immune system dysfunction. Preliminary data and previous literature suggest that autoimmune diseases, and in particular their treatment, may favour the evolution to severe forms of dengue.

Our research hypothesis is that the clinico-biological presentation of dengue might be different in case of autoimmune disease, either on the side of overactivation (autoimmune and auto inflammatory diseases without treatment) or immunodepression (autoimmune and auto inflammatory diseases under immunosuppressive treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient with autoimmune or autoinflammatory disease
* Confirmed diagnosis of dengue (in 2020 or 2021): serological test, antigenic test or PCR test to confirm the diagnosis according to current criteria

Exclusion Criteria:

* minor
* opposition to the re-use of data
* patient not followed in Reunion
* protected adult (guardianship or curatorship) or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic autoimmune disease who have contracted a proven episode of dengue in 2020-21. Only patients followed up at the University Hospital of La Reunion or the Centre Hospitalier Ouest Reunion (CHOR), with or without immunosuppressive treatment will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To assess the observed severity of dengue in patients with autoimmune/autoinflammatory diseases. | Day 1
  Proportion of severe dengue (WHO 2009 definition) in patients with autoimmune/autoinflammatory disease who contracted dengue in 2020/2021, with 95% confidence interval (CI95%).

CONTACTS AND LOCATIONS:
Overall Officials: Loïc RAFFRAY, MD, Principal Investigator — CHU de la Réunion

IPD SHARING:
Plan to Share IPD: No